CLINICAL TRIAL: NCT03910036
Title: Does Post-Operative Intra-Articular Platelet Rich Plasma Injection Improve Meniscal Repair Outcomes
Brief Title: Effect of PRP Injection After Arthroscopic Meniscal Repair in the Healing Process
Acronym: KneePRP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Collaborators: University of Alexandria (Other)
Responsible Party: Principal Investigator, Rehab Abdelaal ELnemr, lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0303544
Record Dates: First submitted 2019-04-06; First posted 2019-04-10 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Knee Pain; Knee Injuries
Keywords: PRP; regeneration; ultrasound
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Intervention Model Description: The study was done on 30 patients underwent arthroscopic isolated meniscal repairs performed by a single surgeon but unfortunately didn't receive PRP injection during the repair procedure. Pre-injection guidelines were given to all patients (in PRP group) in the form of stopping steroidal and non-steroidal anti-inflammatory drugs for at least one week before the procedure, as well as stopping any anticoagulant drugs 5 days before the procedure, increasing intake of fluids within the 24 hours prior to the procedure and anti-anxiety medication were required for anxious patients. Injection, under complete aseptic techniques, was performed while the patient was in supine position, and the knee was fully extended, using the lateral approach. Patients were instructed after injection to avoid using the injected leg for 24 hours, to use ice packs over the injected joint and not to use NSAIDs for another one week.
Who Masked: Outcomes Assessor
Masking Description: the outcome measures assessors were blinded to subjects who receive injection and those who didn't
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PRP group (Experimental): 15 patients to constitute the PRP-group was injected intra-articularly with about 5 ml of PRP in the operated knee joint
  Interventions: Biological: platelet rich plasma
- control group (No Intervention): The other fifteen patients were not injected and constituted control group.

INTERVENTIONS:
Biological: platelet rich plasma — Thirty ml of venous blood was taken from every patient and collected in sodium citrated sterile tubes. Platelet concentrates obtained by adjusting centrifuge at 1800 rpm for 15 min to separate erythrocytes, then at 3500 rpm for 10 min to concentrate the platelets. The preparation was done by a single laboratory technician. Thus 5 ml of PRP were obtained, 0.2 mL of 10% calcium chloride was added to the final product to activate the platelets and injected immediately without storage.
  Arms: PRP group

SUMMARY:
The investigator's hypothesis was that intra-articular knee injection with PRP in patients underwent arthroscopic meniscal repair and didn't receive intra-surgical PRP, may add beneficial effect on post-meniscal repair outcomes regarding pain, functional state of the operated knee as well as healing process.

DETAILED DESCRIPTION:
The study was done on 30 patients underwent arthroscopic isolated meniscal repairs performed by a single surgeon but unfortunately didn't receive PRP injection during the repair procedure.

Random, double blinded selection of 15 patients to constitute the PRP-group was injected intra-articularly with about 5 ml of PRP in the operated knee joint. The other fifteen patients were not injected and constituted control group. PRP preparation:

Thirty ml of venous blood was taken from every patient and collected in sodium citrated sterile tubes. Platelet concentrates obtained by adjusting centrifuge at 1800 rpm for 15 min to separate erythrocytes, then at 3500 rpm for 10 min to concentrate the platelets. The preparation was done by a single laboratory technician. Thus 5 ml of PRP were obtained, 0.2 mL of 10% calcium chloride was added to the final product to activate the platelets and injected immediately without storage. Procedure Pre-injection guidelines were given to all patients (in PRP group) in the form of stopping steroidal and non-steroidal anti-inflammatory drugs for at least one week before the procedure, as well as stopping any anticoagulant drugs 5 days before the procedure, increasing intake of fluids within the 24 hours prior to the procedure and anti-anxiety medication were required for anxious patients. Injection, under complete aseptic techniques, was performed while the patient was in supine position, and the knee was fully extended, using the lateral approach. Patients were instructed after injection to avoid using the injected leg for 24 hours, to use ice packs over the injected joint and not to use NSAIDs for another one week.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-55 years
* Complete meniscal tear in red-white zone done repaired
* Surgery was done by by a single surgeon

Exclusion Criteria:

* Some systemic disorders, such as diabetes, autoimmune diseases, hematological disorders, cardiovascular diseases, infections
* Local knee injuries other than meniscal injury
* Patients receiving treatment with anticoagulants-anti-aggregates
* Use of NSAIDs within 5 days before local PRP injection.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
knee Pain | 3 months
  visual analogue scale, a line 10cm long, zero represent no pain and 10 represent maximal pain, the patient is asked to put a mark that describe his pain
Knee function | 3 months
  Knee injury and osteoarthritis outcome score, assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life. The KOOS's five patient-relevant dimensions are scored separately: Pain (nine items); Symptoms (seven items); ADL Function (17 items); Sport and Recreation Function (five items); Quality of Life (four items). A Likert scale is used and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems
meniscal healing process | 3 months
  by ultrasonography

SECONDARY OUTCOMES:
knee pain | 6 months
  visual analogue scale, a line 10cm long, zero represent no pain and 10 represent maximal pain, the patient is asked to put a mark that describe his pain
knee function | 6 months
  Knee injury and osteoarthritis outcome score, assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life. The KOOS's five patient-relevant dimensions are scored separately: Pain (nine items); Symptoms (seven items); ADL Function (17 items); Sport and Recreation Function (five items); Quality of Life (four items). A Likert scale is used and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems
meniscal healing | 6 months
  by ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Rehab A ELnemr, lecturer, Principal Investigator — Alexandria University, faculty of medicine
Locations (1):
- Rehab Abdelaal ELnemr, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No